CLINICAL TRIAL: NCT03343951
Title: Clinical Examination by Extended Scope Physiotherapists and Orthopaedic Surgeons in an Outpatient Shoulder Clinic: Agreement on Diagnosis and Treatment Plan and Evaluation of Costs and Organisation
Brief Title: Evaluation of Extended Scope Physiotherapists in an Orthopaedic Outpatient Shoulder Clinic
Status: Completed | Type: Observational
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 654821
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-02

CONDITIONS: Shoulder Injuries and Disorders; Shoulder Pain; Musculoskeletal Pain
Keywords: Physical Therapists; Diagnosis; Clinical Competence; Interprofessional Relations; Cost Analysis
MeSH Terms: conditions — Shoulder Injuries; Disease; Shoulder Pain; Musculoskeletal Pain | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Shoulder patients: Shoulder patients referred to examination at the shoulder clinic, Silkeborg Regional Hospital.
  Interventions: Other: Examination

INTERVENTIONS:
Other: Examination — Patients will be examined twice the same day by an extended scope physiotherapist (ESP) and an orthopaedic surgeon (OS) in random order. They will independently and blinded to each other's opinion register
  * diagnosis and treatment plan (including need for further diagnostic examinations - i.e. imaging)
  * if the patient needs a new appointment at the shoulder clinic
  * if they under usual conditions would discuss their results with the opposite health professional before deciding diagnosis and treatment plan.
  After the individual examinations the ESP and OS discuss their results and come to an agreement (common decision) regarding the patient's diagnosis, treatment plan and need of a new appointment. Patients will be informed only of the common decision of the ESP and OS.

SUMMARY:
This study investigates the agreement between extended scope physiotherapists (ESP) and orthopaedic surgeons (OS) on diagnosis and treatment plan in an orthopaedic outpatient shoulder clinic. Furthermore a cost analysis and an evaluation of the interdisciplinary collaboration at the orthopaedic outpatient shoulder clinic (termed shoulder clinic in the following) will be performed.

DETAILED DESCRIPTION:
According to current practice, patients referred from a general practitioner (GP) to the Orthopaedic Outpatient Shoulder Clinic, Silkeborg Regional Hospital (SRH), Denmark, will be examined by either an orthopaedic surgeon (OS) or an extended scope physiotherapist (ESP), as these two groups of health professionals share this assignment. The decision on, which health professional is considered most appropriate to examine the patient, is done by a senior orthopaedic surgeon based on the available information in the referral letter from the GP. Three categories of appropriateness are used: most appropriate to be examined by an OS, most appropriate to be examined by an ESP and equally appropriate to be examined by an ESP or an OS.

The overall purpose of this study is to evaluate the quality of the shared assignment investigated through both professional and organisational outcomes. The following three subsidiary objectives are used:

1. To estimate the agreement between ESP's and OS's on diagnosis and treatment plan (primary subsidiary objective)
2. To estimate direct hospital costs of an examination performed by an ESP and an OS, respectively, and to estimate the difference in costs.
3. To describe the interdisciplinary collaborative practice including evaluation of the extent of relational coordination.

Methods are described underneath related to each subsidiary objective.

1. The study is conducted at the shoulder clinic, SRH. Eligibility criteria, intervention and outcomes are described elsewhere.

   Primary analysis:

   Agreement between ESP and OS in choice of treatment plan (three categories: 1) referral to physiotherapy, 2) need of further diagnostic examination, steroid injection or surgery and 3) no intervention) will be evaluated by estimating the proportion of agreement between
   * The individual registrations of the ESP and OS
   * The individual registration of the ESP and the common decision
   * The individual registration of the OS and the common decision Furthermore, McNemar's test will be used to compare the individual registrations of the ESP and OS, respectively, against the common decision

   Secondary analyses:

   Agreement between ESP and OS in choice of treatment plan (five categories: as described in the outcome section) will be evaluated the same way as described above.

   Agreement between ESP and OS in diagnosis of the patient will be evaluated by estimating both the proportion of total agreement and partial agreement between the two health professionals. Total agreement is defined as ESP and OS having registered the same primary diagnosis. Partial agreement is defined as ESP and OS having registered the same diagnosis but one of them considers it the primary diagnosis while the other considers it a secondary diagnosis.
2. Mean hospital costs of an examination of a shoulder patient will be estimated based on the cohort used to evaluate agreement on diagnosis and treatment plan. Mean hospital costs per patient in the cohort will be estimated separately for ESP's and OS's based on salaries for the health professionals and amount of ordered supplemental diagnostic examinations (X-ray, MR imaging, MR arthrography, CT imaging, ENG, EMG) in each group. Difference in costs will be estimated.
3. Relational coordination in interdisciplinary collaborative practice will be described through separate semi-structured group interviews with ESP's and OS's, respectively.

The Association of Danish Physiotherapists is partly funding the salary for the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18 years
* Referred to The Shoulder Clinic at Silkeborg Regional Hospital
* Considered equally appropriate to be examined by an ESP or an OS
* Ability to read and understand Danish

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with shoulder problems referred to the shoulder clinic at Silkeborg Regional Hospital.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Treatment plan - orthopaedic surgeon | Baseline
  Treatment plan suggested by the OS will be registered in a chart developed for the occasion. The chart has 5 pre-defined categories: 1) referral to physiotherapy, 2) referral to diagnostic examination, 3) steroid injection, 4) surgery and 5) no intervention (categorical)
Treatment plan - physiotherapist | Baseline
  Treatment plan suggested by the ESP will be registered in a chart developed for the occasion. The chart has the same 5 pre-defined categories as for the OS: 1) referral to physiotherapy, 2) referral to diagnostic examination, 3) steroid injection, 4) surgery and 5) no intervention (categorical)
Treatment plan - common decision | Baseline
  The OS and ESP will discuss their results until they agree which treatment plan to offer the patient. Their decision will be registered in a chart developed for the occasion. The chart has the same 5 pre-defined categories as for the individual examinations: 1) referral to physiotherapy, 2) referral to diagnostic examination, 3) steroid injection, 4) surgery and 5) no intervention (categorical)

SECONDARY OUTCOMES:
Diagnosis - orthopaedic surgeon | Baseline
  One primary diagnosis (and if relevant secondary diagnoses) suggested by the OS will be registered in a chart developed for the occasion. The chart has 9 pre-defined categories of diagnoses: 1) impingement, 2) rotator cuff injury, 3) glenohumeral instability, 4) glenohumeral osteoarthritis, 5) periarthritis humeroscapularis, 6) scapular instability, 7) fracture sequelae, 8) acromioclavicular joint disorder, 9) non-related shoulder diagnoses (categorical).
Diagnosis - physiotherapist | Baseline
  One primary diagnosis (and if relevant secondary diagnoses) suggested by the ESP will be registered in a chart developed for the occasion. The chart has the same 9 pre-defined categories of diagnoses as for the OS (categorical).
Diagnosis - common decision | Baseline
  The OS and ESP will discuss their results until they agree on patient diagnosis. Their decision will be registered in a chart developed for the occasion. The chart has the same 9 pre-defined categories of diagnoses as for the individual examinations (categorical).
New appointment - orthopaedic surgeon | Baseline
  The OS registers whether he considers, that the patient should be offered a new appointment at the shoulder clinic (categorical, yes/no)
New appointment - physiotherapist | Baseline
  The ESP registers whether he/she considers, that the patient should be offered a new appointment at the shoulder clinic (categorical, yes/no)
New appointment - common decision | Baseline
  The OS and ESP will discuss their results until they agree, whether the patient should have a new appointment at the shoulder clinic or not. Their decision will be registered (categorical, yes/no)
Discussion needed - orthopaedic surgeon | Baseline
  The OS registers whether he under usual conditions would discuss his results with an ESP before making a decision on diagnosis or treatment plan (categorical, yes/no).
Discussion needed - physiotherapist | Baseline
  The ESP registers whether he/she under usual conditions would discuss his/her results with an OS before making a decision on diagnosis or treatment plan (categorical, yes/no).

OTHER OUTCOMES:
Salary - orthopaedic surgeon, first clinical examination | Baseline
  Mean expenditure on salary for an OS performing a clinical examination of a shoulder patient at the first visit. The estimate will be calculated based on time spent on the examination and mean salary for an OS (information on mean salary will be obtained from statistics at the finance department at the hospital)
Salary - orthopaedic surgeon, planned new appointment | Baseline
  Mean expenditure on salary for an OS performing a follow up appointment with a shoulder patient. The estimate will be calculated based on time spent on the appointment and mean salary for an OS (information on mean salary will be obtained from statistics at the finance department at the hospital)
Salary - extended scope physiotherapist, first clinical examination | Baseline
  Mean expenditure on salary for an ESP performing a clinical examination of a shoulder patient at the first visit. The estimate will be calculated based on time spent on the examination and mean salary for an ESP (information on mean salary will be obtained from statistics at the finance department at the hospital)
Salary - extended scope physiotherapist, planned new appointment | Baseline
  Mean expenditure on salary for an ESP performing a follow up appointment with a shoulder patient. The estimate will be calculated based on time spent on the appointment and mean salary for an ESP (information on mean salary will be obtained from statistics at the finance department at the hospital)
Costs - computed tomography (CT) imaging | Baseline
  Expenditure on CT imaging. Estimate obtained from the finance department at the hospital.
Costs - magnetic resonance (MR) imaging | Baseline
  Expenditure on MR imaging. Estimate obtained from the finance department at the hospital.
Costs - MR arthrography | Baseline
  Expenditure on MR arthrography. Estimate obtained from the finance department at the hospital.
Costs - electroneurography (ENG) | Baseline
  Expenditure on ENG. Estimate obtained from the finance department at the hospital.
Costs - electromyography (EMG) | Baseline
  Expenditure on EMG. Estimate obtained from the finance department at the hospital.
Costs - X-ray | Baseline
  Expenditure on X-ray. Estimate obtained from the finance department at the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Merete N Madsen, MSc, Principal Investigator — Silkeborg Regional Hospital
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madsen MN, Kirkegaard ML, Klebe TM, Linnebjerg CL, Villumsen SMR, Due SJ, Trostrup J, Rossen CB, Birk HO, Elmengaard B, Mikkelsen LR. Inter-professional agreement and collaboration between extended scope physiotherapists and orthopaedic surgeons in an orthopaedic outpatient shoulder clinic - a mixed methods study. BMC Musculoskelet Disord. 2021 Jan 4;22(1):4. doi: 10.1186/s12891-020-03831-z. PMID 33397350